CLINICAL TRIAL: NCT01329419
Title: A Post-marketing Surveillance to Monitor the Safety of HEPSERA(Adefovir Dipivoxil 10mg) Adminstered in Korean Subjects According to the Prescribing Information
Brief Title: HEPSERA Post Marketing Surveillance
Acronym: HEPSERA PMS
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 105711
Record Dates: First submitted 2011-03-10; First posted 2011-04-05 (Estimated); Results first posted 2011-04-05 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — adefovir dipivoxil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- adefovir dipivoxil: Patients administrated adefovir at the site
  Interventions: Drug: adefovir dipivoxil

INTERVENTIONS:
Drug: adefovir dipivoxil — Basically there is no treatment allocation. Subjects who would be administered of adefovir at their physicians' discretion will be enrolled. Dosage regimen will be recommended according to the prescribing information. Subjects will be enrolled consecutively.

SUMMARY:
An open label, multi-centre, non-interventional post-marketing surveillance to monitor the safety and/or efficacy of adefovir dipivoxil administered in Korean CHB patients according to the prescribing information

DETAILED DESCRIPTION:
This study is a post-marketing surveillance to monitor safety and efficacy of adefovir dipivoxil and identify SAEs, adverse drug reactions (ADRs), and unexpected AEs not described as precautions or warnings and to identify possible factors that have an effect on the AEs and to assess effectiveness of adefovir dipivoxil in real clinical practices after marketing. The subjects are patients prescribed for adefovir dipivoxil by the investigators at the sites based on prescription information in normal clinical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients administrated adefovir dipivoxil at the site

Exclusion Criteria:

* Patients administrated adefovir dipivoxil before center initiated date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients administrated adefovir dipivoxil at the site
Sampling Method: Probability Sample
Enrollment: 4393 (Actual)
Dates: Start 2004-08; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective of this post-marketing surveillance (PMS) study was to monitor the safety and efficacy of Hepsera in the real clinical setting after launch.
Groups:
- Hepsera 10 mg Once a Day: Hepsera tablet containing 10 milligrams (mg) of adefovir dipivoxil administered once daily
Period: Overall Study
Arm/Group | Hepsera 10 mg Once a Day
Started | 4393
Completed | 4158
Not Completed | 235
Not completed — Protocol Violation | 235

BASELINE CHARACTERISTICS:
Arm/Group | Hepsera 10 mg Once a Day
Number analyzed (Participants) | 4158
Age, Continuous [Mean (Standard Deviation); unit: Years] — Baseline characteristics were collected in members of the Intent-to-Treat (ITT) Population, comprised of all participants who had been administered the investigational drug at least once and had undergone all safety assessments.
  Years | 43.9 (11)
Sex/Gender, Customized [Number; unit: Participants] — Baseline characteristics were collected in members of the ITT Population, comprised of all participants who had been administered the investigational drug at least once and had undergone all safety assessments.
  Participants
    Female | 874
    Male | 3280
    Missing | 4
Race/Ethnicity, Customized [Number; unit: participants] — Baseline characteristics were collected in members of the ITT Population, comprised of all participants who had been administered the investigational drug at least once and had undergone all safety assessments.
  participants
    Korean | 4158
    Not Korean | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. For a list of all adverse events occurring during the course of the study, please see the table entitled "Other (non-serious) adverse events" in the Adverse Event section of the results record.
Time Frame: 12 weeks
Population: Intent-to-Treat (ITT) Population: all participants who had been administered the investigational drug at least once and had undergone all safety assessments
Measure: Number; unit: participants
Arm/Group | Hepsera 10 mg Once a Day
Number analyzed (Participants) | 4158
participants | 74

2. Secondary Outcome: Number of Participants With a Serious Adverse Event
Description: A serious adverse event is any untoward medical occurrence that, at any dose: results in death /is life-threatening; requires hospitalization or prolongation of exixting hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or is another medically significant event. For a list of all serious adverse events occurring during the course of the study, please see the table entitled "Serious Adverse Events" in the Adverse Event section of the results record.
Time Frame: 12 weeks
Population: ITT Population
Measure: Number; unit: participants
Groups:
- Hepsera 10 mg Once a Day: Hepsera tablet containing 10 mg of adefovir dipivoxil administered once daily
Arm/Group | Hepsera 10 mg Once a Day
Number analyzed (Participants) | 4158
participants | 32

3. Secondary Outcome: Number of Participants With the Indicated Unexpected Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Unexpected adverse events include those not listed in the approved product information and not described as precautions or warnings.
Time Frame: 12 weeks
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Hepsera 10 mg Once a Day
Number analyzed (Participants) | 4158
participants
  Sputum Increased | 5
  Hepatic Cirrhosis | 4
  Hepatic Encephalopathy | 2
  Hepatic Neoplasm | 7
  Hypoaesthesia | 2
  Hemoptysis | 1
  Azotaemia | 1
  Marrow Hyperplasia | 1
  Marrow Depression | 1
  Fracture | 1
  Fasciitis Necrotising | 1
  Skin Reaction Localised | 1
  Myalgia | 1
  Resistance | 1
  Proteinuria | 1
  Edema Peripheral | 1
  Dysuria | 2
  Pancytopenia | 1
  Ascites | 3
  Splenomegaly | 1
  Hernia Inguinal | 1
  Esophageal Varices | 1
  Urethral Disorder | 1
  Erythrocytes Abnormal | 1
  Vein Varicose | 4
  Hemorrhage Rectum | 1
  Gastric Ulcer Hemorrhagic | 1
  Hematemesis | 1
  Pneumonia | 2
  Pulmonary Carcinoma | 1
  Fatigue | 3
  Dyspnea | 1
  Jaundice | 2
  Melaena | 1

ADVERSE EVENTS:
Time Frame: February 19, 2004 to February 18, 2010
Description: Adverse events were coded by using World Health Organization Adverse Reactions Terminology (WHOART, preferred term level) according to the local regulation.
Arm/Group | Hepsera 10 mg Once a Day
Serious Adverse Events (participants affected / at risk) | 32/4158
Other Adverse Events (participants affected / at risk) | 74/4158
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hepsera 10 mg Once a Day (N=4158)
Hepatic Failure (Hepatobiliary disorders) | 9
Hepatic Cirrhosis (Hepatobiliary disorders) | 4
Vein Varicose (Blood and lymphatic system disorders) | 3
Gastric Ulcer Hemorrhagic (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Hematemesis (Gastrointestinal disorders) | 1
Hypoaesthesia (Nervous system disorders) | 1
Hepatic Encephalopathy (Hepatobiliary disorders) | 2
Abdominal Pain (Gastrointestinal disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Jaundice (Hepatobiliary disorders) | 2
Alanine Transaminase/Aspartate Aminotransferase Increased (Hepatobiliary disorders) | 1
Fever (General disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Ascites (General disorders) | 1
Pulmonary Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Fracture (Musculoskeletal and connective tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Hernia Inguinal (Reproductive system and breast disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Fasciitis Necrotising (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Hepsera 10 mg Once a Day (N=4158)
Abdominal Pain (Gastrointestinal disorders) | 6
Dyspepsia (Gastrointestinal disorders) | 5
Gagging (Gastrointestinal disorders) | 4
Flatulence (Gastrointestinal disorders) | 4
Diarrhea (General disorders) | 2
Esophageal Varices (Gastrointestinal disorders) | 1
Hemorrhage Rectum (Gastrointestinal disorders) | 1
Gastric Ulcer Hemorrhagic (Gastrointestinal disorders) | 1
Hematemesis (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 1
Hepatic Failure (Hepatobiliary disorders) | 9
Hepatic Cirrhosis (Hepatobiliary disorders) | 4
Alanine Transaminase/Aspartate Aminotransferase Increased (Hepatobiliary disorders) | 2
Hepatic Encephalopathy (Hepatobiliary disorders) | 2
Hepatitis Chronic Active Aggrava (Hepatobiliary disorders) | 2
Jaundice (Hepatobiliary disorders) | 2
Asthenia (General disorders) | 5
Ascites (General disorders) | 3
Fatigue (General disorders) | 3
Tolerance (General disorders) | 1
Edema Peripheral (General disorders) | 1
Fever (General disorders) | 1
Coughing (Respiratory, thoracic and mediastinal disorders) | 7
Sputum Increased (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Hepatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7
Pulmonary Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysuria (Renal and urinary disorders) | 2
Azotaemia (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Urethral Disorder (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin Reaction Localised (Skin and subcutaneous tissue disorders) | 1
Vein Varicose (Blood and lymphatic system disorders) | 4
Fracture (Musculoskeletal and connective tissue disorders) | 1
Fasciitis Necrotising (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Headache (Nervous system disorders) | 1
Hernia Inguinal (Renal and urinary disorders) | 1
Red Blood Cell Abnormality (Blood and lymphatic system disorders) | 1
Marrow Hyperplasia (Blood and lymphatic system disorders) | 1
Marrow Depression (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Splenomegaly (Blood and lymphatic system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.